CLINICAL TRIAL: NCT02656303
Title: A Multi-Center, Open-Label, Compassionate Use Extension Study of Ublituximab (TG-1101) in Combination With Umbralisib (TGR-1202) for Patients Previously Enrolled in Protocol UTX-TGR-304
Brief Title: A Study to Evaluate the Safety and Efficacy of Ublituximab in Combination With Umbralisib for Participants Previously Enrolled in Protocol UTX-TGR-304
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Strategic/Business Decision
Sponsor: TG Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UTX-TGR-204; 2016-004339-19 (EudraCT Number)
Record Dates: First submitted 2016-01-13; First posted 2016-01-14 (Estimated); Results first posted 2023-06-22 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-05

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ublituximab; umbralisib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Parent Study Arm B (Experimental): Participants from Arm B of the parent trial (UTX-TGR-304) received ublituximab, 150 milligrams (mg), intravenously (IV), on Day 1, 750 mg on Day 2, followed by 900 mg on Days 8 and 15 of Cycle 1 (cycle length=28 days), Day 1 of Cycles 2-6, and once every 3 months thereafter, along with umbralisib, 800 mg, orally, once daily during each cycle until disease progression, lack of tolerability, or until the treatment is commercially available or up to 78 months.
  Interventions: Biological: Ublituximab; Drug: Umbralisib
- Parent Study Arm C (Experimental): Participants from Arm C of the parent trial (UTX-TGR-304) received ublituximab, 900 mg, IV, on Day 1 of Cycles 1-6 (cycle length=28 days), and once every 3 months thereafter, along with umbralisib, 800 mg, orally, once daily during each cycle until disease progression, lack of tolerability, or until the treatment is commercially available or up to 78 months.
  Interventions: Biological: Ublituximab; Drug: Umbralisib
- Parent Study Arm D (Experimental): Participants from Arm D of the parent trial (UTX-TGR-304) received ublituximab, 150 mg, IV, on Day 1, 750 mg on Day 2, followed by 900 mg on Days 8 and 15 of Cycle 1 (cycle length=28 days), Day 1 of Cycles 2-6, and once every 3 months thereafter, along with umbralisib, 800 mg, orally, once daily during each cycle until disease progression, lack of tolerability, or until the treatment is commercially available or up to 78 months.
  Interventions: Biological: Ublituximab; Drug: Umbralisib

INTERVENTIONS:
Biological: Ublituximab — Ublituximab IV infusion
  Other Names: TG-1101
Drug: Umbralisib — Umbralisib tablets
  Other Names: TGR-1202

SUMMARY:
The purpose of this study was to provide the opportunity to the participants who progressed on treatment arm previously in the study UTX-TGR-304 (NCT02612311) to receive ublituximab (TG-1101) treatment in combination with umbralisib (TGR-1202).

ELIGIBILITY:
Inclusion Criteria:

* Prior treatment in clinical trial UTX-TGR-304
* Eastern Cooperative Oncology Group (ECOG) score of 0 to 2

Exclusion Criteria:

* Participants refractory to ublituximab + TGR-1202
* Transformation of chronic lymphocytic leukemia (CLL) to aggressive Non-Hodgkin's Lymphoma (NHL) (Richter's transformation)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2016-01-07 (Actual); Primary Completion 2022-05-26 (Actual); Study Completion 2022-07-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (80):
- United States (66):
  - TG Therapeutics Investigational Trial Site, Huntsville, Alabama
  - TG Therapeutics Investigational Trial Site, Chandler, Arizona
  - TG Therapeutics Investigational Trial Site, Fayetteville, Arkansas
  - TG Therapeutics Investigational Trial Site, Duarte, California
  - TG Therapeutics Investigational Trial Site, Pleasanton, California
  - TG Therapeutics Investigational Trial Site, San Diego, California
  - TG Therapeutics Investigational Trial Site, Whittier, California
  - TG Therapeutics Investigational Trial Site, Aurora, Colorado
  - TG Therapeutics Investigational Trial Site, Denver, Colorado
  - TG Therapeutics Investigational Trial Site, Bridgeport, Connecticut
  - TG Therapeutics Investigational Trial Site, New Haven, Connecticut
  - TG Therapeutics Investigational Trial Site, Stamford, Connecticut
  - TG Therapeutics Investigational Trial Site, Newark, Delaware
  - TG Therapeutics Investigational Trial Site, Boca Raton, Florida
  - TG Therapeutics Investigational Trial Site, Fort Myers, Florida
  - TG Therapeutics Investigational Trial Site, Jacksonville, Florida
  - TG Therapeutics Investigational Trial Site, St. Petersburg, Florida
  - TG Therapeutics Investigational Trial Site, Tallahassee, Florida
  - TG Therapeutics Investigational Trial Site, West Palm Beach, Florida
  - TG Therapeutics Investigational Trial Site, Albany, Georgia
  - TG Therapeutics Investigational Trial Site, Chicago, Illinois
  - TG Therapeutics Investigational Trial Site, Peoria, Illinois
  - TG Therapeutics Investigational Trial Site, Swansea, Illinois
  - TG Therapeutics Investigational Trial Site, Urbana, Illinois
  - TG Therapeutics Investigational Trial Site, Fort Wayne, Indiana
  - TG Therapeutics Investigational Trial Site, Indianapolis, Indiana
  - TG Therapeutics Investigational Trial Site, Westwood, Kansas
  - TG Therapeutics Investigational Trial Site, Louisville, Kentucky
  - TG Therapeutics Investigational Trial Site, Worcester, Massachusetts
  - TG Therapeutics Investigational Trial Site, Ann Arbor, Michigan
  - TG Therapeutics Investigational Trial Site, Detroit, Michigan
  - TG Therapeutics Investigational Trial Site, Jackson, Michigan
  - TG Therapeutics Investigational Trial Site, Saint Louis Park, Minnesota
  - TG Therapeutics Investigational Trial Site, Kansas City, Missouri
  - TG Therapeutics Investigational Trial Site, Lincoln, Nebraska
  - TG Therapeutics Investigational Trial Site, Lebanon, New Hampshire
  - TG Therapeutics Investigational Trial Site, Morristown, New Jersey
  - TG Therapeutics Investigational Trial Site, Glens Falls, New York
  - TG Therapeutics Investigational Trial Site, Syracuse, New York
  - TG Therapeutics Investigational Trial Site, Charlotte, North Carolina
  - TG Therapeutics Investigational Trial Site, Durham, North Carolina
  - TG Therapeutics Investigational Trial Site, Hickory, North Carolina
  - TG Therapeutics Investigational Trial Site, Kinston, North Carolina
  - TG Therapeutics Investigational Trial Site, Washington, North Carolina
  - TG Therapeutics Investigational Trial Site, Canton, Ohio
  - TG Therapeutics Investigational Trial Site, Toledo, Ohio
  - TG Therapeutics Investigational Trial Site, Portland, Oregon
  - TG Therapeutics Investigational Trial Site, Springfield, Oregon
  - TG Therapeutics Investigational Trial Site, Camp Hill, Pennsylvania
  - TG Therapeutics Investigational Trial Site, Hershey, Pennsylvania
  - TG Therapeutics Investigational Trial Site, Philadelphia, Pennsylvania
  - TG Therapeutics Investigational Trial Site, Pittsburgh, Pennsylvania
  - TG Therapeutics Investigational Trial Site, Pawtucket, Rhode Island
  - TG Therapeutics Investigational Trial Site, Greenville, South Carolina
  - TG Therapeutics Investigational Trial Site, Sioux Falls, South Dakota
  - TG Therapeutics Investigational Trial Site, Chattanooga, Tennessee
  - TG Therapeutics Investigational Trial Site, Nashville, Tennessee
  - TG Therapeutics Investigational Trial Site, Fort Worth, Texas
  - TG Therapeutics Investigational Trial Site, San Antonio, Texas
  - TG Therapeutics Investigational Trial Site, Ogden, Utah
  - TG Therapeutics Investigational Trial Site, Blacksburg, Virginia
  - TG Therapeutics Investigational Trial Site, Charlottesville, Virginia
  - TG Therapeutics Investigational Trial Site, Fort Belvoir, Virginia
  - TG Therapeutics Investigational Trial Site, Seattle, Washington
  - TG Therapeutics Investigational Trial Site, Spokane, Washington
  - TG Therapeutics Investigational Trial Site, Wauwatosa, Wisconsin
- Italy (3):
  - TG Therapeutics Investigational Trial Site, Ferrara
  - TG Therapeutics Investigational Trial Site, Milan
  - TG Therapeutics Investigational Trial Site, Torino
- Poland (7):
  - TG Therapeutics Investigational Trial Site, Chorzów
  - TG Therapeutics Investigational Trial Site, Gdynia
  - TG Therapeutics Investigational Trial Site, Krakow
  - TG Therapeutics Investigational Trial Site, Lodz
  - TG Therapeutics Investigational Trial Site, Lublin
  - TG Therapeutics Investigational Trial Site, Słupsk
  - TG Therapeutics Investigational Trial Site, Warsaw
- United Kingdom (4):
  - TG Therapeutics Investigational Trial Site, London
  - TG Therapeutics Investigational Trial Site, Norwich
  - TG Therapeutics Investigational Trial Site, Sunderland
  - TG Therapeutics Investigational Trial Site, Wolverhampton

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 116 participants took part across 50 investigative sites in the United States, United Kingdom, Italy, and Poland from 07 January 2016 to 11 July 2022.
Period: Overall Study
Arm/Group | Parent Study Arm B | Parent Study Arm C | Parent Study Arm D
Started | 67 | 31 | 18
Completed | 0 | 0 | 0
Not Completed | 67 | 31 | 18
Not completed — Adverse Event | 3 | 2 | 0
Not completed — Death | 12 | 4 | 1
Not completed — Lack of Efficacy | 1 | 0 | 0
Not completed — Non-Compliance with Study | 1 | 1 | 0
Not completed — Investigator Decision | 2 | 1 | 0
Not completed — Progressive Disease | 25 | 14 | 10
Not completed — Study Terminated by Sponsor | 20 | 7 | 5
Not completed — Withdrawal of Consent by Participants | 1 | 1 | 0
Not completed — Initiation of Non-protocol Intervention | 1 | 0 | 0
Not completed — Reason not Specified | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Population: The Safety Population included all participants who were enrolled and received at least one dose of study drug.
Groups:
- Parent Study Arm B: Participants from Arm B of the parent trial (UTX-TGR-304) received ublituximab, 150 mg, IV, on Day 1, 750 mg on Day 2, followed by 900 mg on Days 8 and 15 of Cycle 1 (cycle length=28 days), Day 1 of Cycles 2-6, and once every 3 months thereafter, along with umbralisib, 800 mg, orally, once daily during each cycle until disease progression, lack of tolerability, or until the treatment is commercially available or up to 78 months.
- Total: Total of all reporting groups
Arm/Group | Parent Study Arm B | Parent Study Arm C | Parent Study Arm D | Total
Number analyzed (Participants) | 67 | 31 | 18 | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.6 (8.18) | 66.7 (9.41) | 65.7 (8.79) | 65.9 (8.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 5 | 5 | 29
  Male | 48 | 26 | 13 | 87
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1 | 2
  Not Hispanic or Latino | 66 | 30 | 16 | 112
  Unknown or Not Reported | 0 | 1 | 1 | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 65 | 30 | 15 | 110
  Race: Black or African American | 2 | 0 | 1 | 3
  Race: Other | 0 | 0 | 2 | 2
  Race: Not Reported | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) as Per International Workshop on Chronic Lymphocytic Leukemia (iwCLL) Criteria
Description: ORR was defined as sum of participants with partial responses (PR) and complete responses (CR). CR: No evidence of new disease; Absolute lymphocyte count(ALC)<4x10^9/liter(L); Regression of all target nodal masses to ≤1.5 centimeters (cm) in longest diameter(LD); Normal spleen,liver size; Regression to normal of all nodal non-target disease and disappearance of all detectable; Non-nodal, non-target disease; Morphologically negative bone marrow; No lymphoid nodules; Absolute neutrophil count(ANC)>1.5x10^9/L,platelets≥100x10^9/L,hemoglobin (Hgb)≥110 gram per liter(g/L). PR: No evidence of new disease; Response in 2 of following if abnormal at baseline: ALC<4x10^9/L or ≥50% decrease from baseline in sum of products(SPD) of target nodal lesions; splenomegaly; hepatomegaly;≥50% decrease from baseline in CLL marrow infiltrate/B-lymphoid nodules; response in any 1:ANC>1.5x10^9/L,platelets>100x10^9/L,Hgb>110g/L or ≥50% increase over baseline in any of these.
Time Frame: Up to 76 months
Population: Data for this outcome measure was not collected or analyzed as the study was terminated due to sponsor's business decision.
Arm/Group | Parent Study Arm B | Parent Study Arm C | Parent Study Arm D
Number analyzed (Participants) | 0 | 0 | 0

2. Primary Outcome: Complete Response (CR) Rate Per iwCLL Criteria
Description: The CR rate was defined as the percentage of participants who achieved CR. CR: No evidence of new disease; ALC <4 x 10^9/L; Regression of all target nodal masses to normal size ≤1.5 cm in the LD; Normal spleen and liver size; Regression to normal of all nodal non-target disease and disappearance of all detectable; Non-nodal, non-target disease; Morphologically negative bone marrow; No lymphoid nodules; ANC >1.5 x 10^9/L, platelets ≥100 x 10^9/L, Hgb ≥110 g/L.
Time Frame: Up to 76 months
Population: as for outcome 1
Arm/Group | Parent Study Arm B | Parent Study Arm C | Parent Study Arm D
Number analyzed (Participants) | 0 | 0 | 0

3. Primary Outcome: Progression-Free Survival (PFS) Per iwCLL Criteria
Description: PFS was defined as the interval from enrollment to the earlier of the first documentation of definitive disease progression (PD) or death from any cause. PD was appearance of new nodes >1.5 cm in the LD and >1.0 in longest perpendicular diameter (LPD), new or recurrent hepatomegaly or splenomegaly, new or reappearance of an unequivocal extra-nodal lesion, ≥50% increase from the nadir in the sum of products of diameters (SPD) of target lesions, ≥50% increase in the LD of an individual node or extra-nodal mass, splenic/hepatic enlargement of ≥50% from nadir, unequivocal increase in the size of non-target disease, transformation to a more aggressive histology, decrease in platelet count or Hgb, >50% decrease from the highest on-study platelet count, >20 g/L decrease from the highest on-study Hgb.
Time Frame: Up to 76 months
Population: as for outcome 1
Arm/Group | Parent Study Arm B | Parent Study Arm C | Parent Study Arm D
Number analyzed (Participants) | 0 | 0 | 0

4. Primary Outcome: Duration of Response (DOR)
Description: DOR:Interval from first documentation of CR/PR to first documentation of PD or death from any cause.CR:ALC<4x10^9/L;Regression to normal of target nodal masses,nodal non-target disease,and no detectable non-nodal,non-target disease;Normal spleen,liver size;Morphologically negative bone marrow,No lymphoid nodules;ANC>1.5x10^9/L,Platelets≥100x10^9/L,Hgb≥110 g/L.PR:Response in 2 or more:ALC<4x10^9/L, ≥50% drop from baseline in ALC or SPD of target nodal lesions,Hepatosplenomegaly,≥50% decrease from baseline in CLL marrow infiltrate/B-lymphoid nodules;Response in 1 or more:ANC>1.5x10^9/L,Platelets>100x10^9/L,Hgb>110 g/L or ≥50% increase over baseline in any.PD:Response in 1 or more:new nodes,Hepatosplenomegaly,unequivocal extra-nodal lesion;≥50% increase from nadir in SPD of target lesions or LD of node/extra-nodal mass or Splenic/Hepatic size,Unequivocal increase in non-target disease,More aggressive histology;Drop of >50% in platelets/>20g/L in Hgb from highest on-study count.
Time Frame: Up to 76 months
Population: as for outcome 1
Arm/Group | Parent Study Arm B | Parent Study Arm C | Parent Study Arm D
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Minimal Residual Disease (MRD) Negativity Rate
Description: MRD negativity rate is defined as the percentage of participants who are MRD negative. If a participant was determined to be MRD negative by peripheral blood, a bone marrow aspirate was obtained to assess MRD in the bone marrow.
Time Frame: From Cycle 6 until Cycle 15 (cycle length=28 days) (Up to approximately 76 months)
Population: as for outcome 1
Arm/Group | Parent Study Arm B | Parent Study Arm C | Parent Study Arm D
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Number of Participants Experiencing at Least One Treatment-Emergent Adverse Event (TEAE)
Description: An adverse event (AE) is any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product. An AE does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporarily associated with the use of a medicinal product, whether or not considered related to the medicinal product. TEAE is any AE that occur after first dosing of study medication and through the end of the study or through 30 days after the last dose of study treatment, or is considered treatment-related regardless of the start date of the event, or is present before first dosing of study medication but worsens in intensity or the investigator subsequently considers treatment-related.
Time Frame: Up to 78 months
Population: The Safety Population included all participants who were enrolled and received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Parent Study Arm B | Parent Study Arm C | Parent Study Arm D
Number analyzed (Participants) | 67 | 31 | 18
Participants | 66 | 30 | 18

ADVERSE EVENTS:
Time Frame: Up to approximately 78 months
Description: The Safety Population included all participants who were enrolled and received at least one dose of study drug.
Arm/Group | Parent Study Arm B | Parent Study Arm C | Parent Study Arm D
All-Cause Mortality (participants affected / at risk) | 23/67 | 9/31 | 7/18
Serious Adverse Events (participants affected / at risk) | 36/67 | 13/31 | 8/18
Other Adverse Events (participants affected / at risk) | 65/67 | 30/31 | 17/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Parent Study Arm B (N=67) | Parent Study Arm C (N=31) | Parent Study Arm D (N=18)
Anaemia (Blood and lymphatic system disorders) | 2 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 3 | 0 | 0
Lymph node haemorrhage (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 0 | 0
Colitis (Gastrointestinal disorders) | 2 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0
Chest pain (General disorders) | 1 | 0 | 0
Death (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 1 | 0 | 0
Sudden cardiac death (General disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 1 | 0 | 0
Anaphylactic shock (Immune system disorders) | 0 | 1 | 0
Aspergillus infection (Infections and infestations) | 0 | 0 | 1
Babesiosis (Infections and infestations) | 1 | 0 | 0
Bronchitis (Infections and infestations) | 1 | 0 | 0
COVID-19 (Infections and infestations) | 4 | 1 | 2
COVID-19 pneumonia (Infections and infestations) | 5 | 2 | 2
Cytomegalovirus infection (Infections and infestations) | 0 | 1 | 0
Pneumocystis jirovecii pneumonia (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 8 | 2 | 1
Rectal abscess (Infections and infestations) | 0 | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Septic shock (Infections and infestations) | 2 | 0 | 0
Compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 2 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0
Paraparesis (Nervous system disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 1/48 | 0/26 | 0/13
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Parent Study Arm B (N=67) | Parent Study Arm C (N=31) | Parent Study Arm D (N=18)
Anaemia (Blood and lymphatic system disorders) | 8 | 3 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1 | 0 | 0
Increased tendency to bruise (Blood and lymphatic system disorders) | 1 | 0 | 0
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 1 | 0
Leukocytosis (Blood and lymphatic system disorders) | 1 | 0 | 0
Lymphocytosis (Blood and lymphatic system disorders) | 0 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 17 | 6 | 6
Thrombocytopenia (Blood and lymphatic system disorders) | 4 | 0 | 2
Angina pectoris (Cardiac disorders) | 0 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 2 | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0
Bradycardia (Cardiac disorders) | 0 | 0 | 1
Cardiac failure chronic (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Tachyarrhythmia (Cardiac disorders) | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 2 | 0
Hydrocele (Congenital, familial and genetic disorders) | 1 | 0 | 0
Deafness (Ear and labyrinth disorders) | 1 | 0 | 0
Deafness bilateral (Ear and labyrinth disorders) | 0 | 1 | 0
Deafness unilateral (Ear and labyrinth disorders) | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 1 | 0
Hyperacusis (Ear and labyrinth disorders) | 1 | 0 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 1
Inner ear inflammation (Ear and labyrinth disorders) | 0 | 1 | 0
Meniere's disease (Ear and labyrinth disorders) | 1 | 0 | 0
Middle ear inflammation (Ear and labyrinth disorders) | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 3 | 0 | 1
Vertigo (Ear and labyrinth disorders) | 0 | 2 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0 | 0
Adrenal insufficiency (Endocrine disorders) | 1 | 0 | 0
Age-related macular degeneration (Eye disorders) | 1 | 0 | 0
Blepharitis (Eye disorders) | 0 | 0 | 1
Chalazion (Eye disorders) | 1 | 0 | 0
Conjunctival haemorrhage (Eye disorders) | 1 | 1 | 0
Dry eye (Eye disorders) | 3 | 0 | 0
Eye irritation (Eye disorders) | 1 | 0 | 0
Eye swelling (Eye disorders) | 1 | 0 | 0
Lacrimation increased (Eye disorders) | 2 | 1 | 0
Ocular hyperaemia (Eye disorders) | 1 | 0 | 0
Vision blurred (Eye disorders) | 3 | 1 | 0
Visual brightness (Eye disorders) | 1 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 5 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 5 | 5 | 0
Abdominal pain lower (Gastrointestinal disorders) | 1 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 4 | 4 | 1
Abdominal tenderness (Gastrointestinal disorders) | 1 | 0 | 0
Colitis (Gastrointestinal disorders) | 2 | 2 | 0
Constipation (Gastrointestinal disorders) | 11 | 4 | 2
Dental caries (Gastrointestinal disorders) | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 35 | 11 | 6
Diverticulum intestinal (Gastrointestinal disorders) | 1 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 2 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 9 | 2 | 2
Dysphagia (Gastrointestinal disorders) | 1 | 0 | 0
Enterovesical fistula (Gastrointestinal disorders) | 0 | 1 | 0
Eructation (Gastrointestinal disorders) | 1 | 0 | 0
Faeces soft (Gastrointestinal disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 4 | 2 | 1
Gastric dilatation (Gastrointestinal disorders) | 1 | 0 | 0
Gastric polyps (Gastrointestinal disorders) | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 3 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 3 | 0
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0
Haemoperitoneum (Gastrointestinal disorders) | 0 | 1 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 1
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 29 | 10 | 5
Oral pain (Gastrointestinal disorders) | 1 | 0 | 0
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 1
Rectal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 3 | 0 | 0
Tongue discomfort (Gastrointestinal disorders) | 1 | 0 | 0
Tongue ulceration (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 11 | 3 | 1
Adverse drug reaction (General disorders) | 0 | 0 | 1
Asthenia (General disorders) | 11 | 4 | 2
Axillary pain (General disorders) | 1 | 0 | 0
Catheter site erythema (General disorders) | 1 | 0 | 0
Chest discomfort (General disorders) | 0 | 0 | 1
Chills (General disorders) | 13 | 3 | 0
Face oedema (General disorders) | 0 | 1 | 0
Fatigue (General disorders) | 23 | 12 | 2
Feeling abnormal (General disorders) | 2 | 0 | 0
Feeling cold (General disorders) | 0 | 1 | 1
Gait disturbance (General disorders) | 1 | 1 | 1
Hypothermia (General disorders) | 1 | 0 | 0
Localised oedema (General disorders) | 1 | 0 | 0
Malaise (General disorders) | 2 | 0 | 0
Non-cardiac chest pain (General disorders) | 2 | 1 | 0
Oedema peripheral (General disorders) | 14 | 6 | 3
Peripheral swelling (General disorders) | 1 | 0 | 0
Pyrexia (General disorders) | 14 | 1 | 4
Secretion discharge (General disorders) | 0 | 0 | 1
Swelling (General disorders) | 1 | 0 | 0
Swelling face (General disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 2 | 0 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 0 | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 0 | 1 | 0
Hypertransaminasaemia (Hepatobiliary disorders) | 1 | 0 | 0
Allergy to arthropod bite (Immune system disorders) | 1 | 0 | 0
Contrast media allergy (Immune system disorders) | 2 | 0 | 0
Hypogammaglobulinaemia (Immune system disorders) | 3 | 2 | 2
Seasonal allergy (Immune system disorders) | 0 | 0 | 1
Body tinea (Infections and infestations) | 0 | 1 | 0
Bronchitis (Infections and infestations) | 4 | 3 | 0
COVID-19 (Infections and infestations) | 5 | 0 | 1
Campylobacter infection (Infections and infestations) | 1 | 0 | 0
Candida infection (Infections and infestations) | 2 | 0 | 0
Chronic sinusitis (Infections and infestations) | 2 | 0 | 1
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0
Conjunctivitis (Infections and infestations) | 1 | 0 | 0
Cystitis (Infections and infestations) | 1 | 0 | 0
Cytomegalovirus infection (Infections and infestations) | 2 | 1 | 2
Cytomegalovirus infection reactivation (Infections and infestations) | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0
Ear infection (Infections and infestations) | 2 | 1 | 1
Epididymitis (Infections and infestations) | 1 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0
Fungal oesophagitis (Infections and infestations) | 1 | 0 | 0
Fungal skin infection (Infections and infestations) | 1 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1
Gingivitis (Infections and infestations) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 3 | 1 | 0
Hordeolum (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 4 | 0 | 0
Laryngitis (Infections and infestations) | 0 | 0 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 0
Mastoiditis (Infections and infestations) | 0 | 1 | 0
Mycobacterium avium complex infection (Infections and infestations) | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 2 | 0
Oral candidiasis (Infections and infestations) | 0 | 0 | 1
Otitis media (Infections and infestations) | 1 | 0 | 0
Pharyngitis streptococcal (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 12 | 1 | 4
Pseudomonas infection (Infections and infestations) | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 3 | 0 | 1
Rhinitis (Infections and infestations) | 2 | 0 | 0
Rhinovirus infection (Infections and infestations) | 1 | 0 | 1
Sepsis (Infections and infestations) | 1 | 0 | 1
Sinusitis (Infections and infestations) | 3 | 1 | 1
Skin infection (Infections and infestations) | 1 | 0 | 0
Tooth abscess (Infections and infestations) | 0 | 1 | 0
Tooth infection (Infections and infestations) | 2 | 0 | 0
Upper respiratory tract infection (Infections and infestations) | 14 | 9 | 4
Urinary tract infection (Infections and infestations) | 5 | 2 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 6 | 2 | 1
Fall (Injury, poisoning and procedural complications) | 4 | 1 | 0
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 15 | 5 | 9
Limb injury (Injury, poisoning and procedural complications) | 1 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 0 | 1 | 0
Skin laceration (Injury, poisoning and procedural complications) | 3 | 1 | 0
Skin wound (Injury, poisoning and procedural complications) | 1 | 0 | 0
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 15 | 6 | 3
Aspartate aminotransferase increased (Investigations) | 15 | 4 | 2
Blood alkaline phosphatase increased (Investigations) | 7 | 0 | 1
Blood bicarbonate decreased (Investigations) | 0 | 1 | 0
Blood bilirubin increased (Investigations) | 3 | 3 | 0
Blood creatinine increased (Investigations) | 6 | 3 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 1 | 1
Blood potassium decreased (Investigations) | 0 | 1 | 1
Blood pressure increased (Investigations) | 1 | 1 | 0
Blood sodium decreased (Investigations) | 1 | 0 | 0
Blood urea increased (Investigations) | 1 | 0 | 0
Blood uric acid increased (Investigations) | 0 | 2 | 0
Blood urine present (Investigations) | 0 | 1 | 0
Cardiac murmur (Investigations) | 2 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 2 | 0 | 0
Glomerular filtration rate decreased (Investigations) | 1 | 0 | 0
Haematocrit increased (Investigations) | 1 | 0 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1
Lymphocyte count decreased (Investigations) | 0 | 2 | 2
Lymphocyte count increased (Investigations) | 3 | 0 | 1
Monocyte percentage decreased (Investigations) | 0 | 1 | 0
Neutrophil count decreased (Investigations) | 3 | 3 | 5
Neutrophil percentage decreased (Investigations) | 0 | 1 | 0
Platelet count decreased (Investigations) | 5 | 2 | 2
Prostatic specific antigen increased (Investigations) | 1 | 0 | 0
SARS-CoV-2 test positive (Investigations) | 1 | 0 | 0
Urine output decreased (Investigations) | 0 | 1 | 0
Weight decreased (Investigations) | 6 | 4 | 2
Weight increased (Investigations) | 1 | 0 | 0
White blood cell count decreased (Investigations) | 3 | 2 | 2
White blood cell count increased (Investigations) | 1 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 10 | 1 | 3
Dehydration (Metabolism and nutrition disorders) | 3 | 2 | 0
Food intolerance (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 4 | 0 | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 4 | 0 | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 0 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 5 | 3 | 0
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 2
Hypokalaemia (Metabolism and nutrition disorders) | 9 | 4 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 3 | 1 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 4 | 2 | 2
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 12 | 4 | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 12 | 2 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 3 | 1 | 1
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint effusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6 | 3 | 0
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscle twitching (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 5 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 4 | 4 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 1 | 3
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Acrochordon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Skin papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Ataxia (Nervous system disorders) | 1 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0
Cognitive disorder (Nervous system disorders) | 0 | 1 | 0
Dementia (Nervous system disorders) | 2 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 1 | 0
Dizziness (Nervous system disorders) | 12 | 2 | 1
Drooling (Nervous system disorders) | 1 | 0 | 0
Dysaesthesia (Nervous system disorders) | 1 | 0 | 0
Dysgeusia (Nervous system disorders) | 3 | 4 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 1
Essential tremor (Nervous system disorders) | 1 | 0 | 0
Head discomfort (Nervous system disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 10 | 2 | 1
Hyperaesthesia (Nervous system disorders) | 1 | 0 | 0
Hypoaesthesia (Nervous system disorders) | 3 | 1 | 2
Memory impairment (Nervous system disorders) | 2 | 1 | 0
Myoclonus (Nervous system disorders) | 1 | 0 | 0
Nervous system disorder (Nervous system disorders) | 1 | 0 | 0
Neuropathy peripheral (Nervous system disorders) | 1 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1
Restless legs syndrome (Nervous system disorders) | 1 | 0 | 0
Sciatica (Nervous system disorders) | 2 | 0 | 0
Seizure (Nervous system disorders) | 1 | 0 | 0
Slow speech (Nervous system disorders) | 0 | 0 | 1
Somnolence (Nervous system disorders) | 3 | 0 | 0
Syncope (Nervous system disorders) | 1 | 0 | 0
Tremor (Nervous system disorders) | 8 | 1 | 0
Abnormal dreams (Psychiatric disorders) | 1 | 0 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0
Anxiety (Psychiatric disorders) | 7 | 3 | 0
Confusional state (Psychiatric disorders) | 6 | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0 | 0
Depression (Psychiatric disorders) | 1 | 1 | 1
Hallucination (Psychiatric disorders) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 16 | 5 | 3
Mental status changes (Psychiatric disorders) | 0 | 0 | 1
Mood altered (Psychiatric disorders) | 0 | 0 | 1
Personality change (Psychiatric disorders) | 1 | 0 | 0
Restlessness (Psychiatric disorders) | 1 | 0 | 0
Somatic symptom disorder (Psychiatric disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 3 | 1 | 0
Chromaturia (Renal and urinary disorders) | 1 | 0 | 0
Chronic kidney disease (Renal and urinary disorders) | 2 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 0
Haematuria (Renal and urinary disorders) | 4 | 0 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 1 | 0
Nocturia (Renal and urinary disorders) | 3 | 0 | 1
Pollakiuria (Renal and urinary disorders) | 3 | 2 | 0
Polyuria (Renal and urinary disorders) | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0
Renal cyst (Renal and urinary disorders) | 1 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 2 | 0 | 0
Urinary retention (Renal and urinary disorders) | 2 | 1 | 0
Urinary tract pain (Renal and urinary disorders) | 1 | 1 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Cervical dysplasia (Reproductive system and breast disorders) | 1 | 0 | 0
Haematospermia (Reproductive system and breast disorders) | 1 | 0 | 0
Pelvic discomfort (Reproductive system and breast disorders) | 1 | 0 | 0
Prostatomegaly (Reproductive system and breast disorders) | 1 | 0 | 0
Testicular oedema (Reproductive system and breast disorders) | 0 | 1 | 0
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 22 | 5 | 3
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 4 | 3
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Increased viscosity of upper respiratory secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Lower respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Lung consolidation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
Lung opacity (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 4 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0
Paranasal sinus discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory tract irritation (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 5 | 2 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Tracheomalacia (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Alopecia areata (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dermal cyst (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 2 | 2 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 2 | 1 | 1
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Ingrowing nail (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Miliaria (Skin and subcutaneous tissue disorders) | 2 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 7 | 2 | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Precancerous skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 4 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 6 | 2 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 3 | 3 | 0
Rash pruritic (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin erosion (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Pleurodesis (Surgical and medical procedures) | 0 | 0 | 1
Aortic stenosis (Vascular disorders) | 2 | 0 | 0
Arteriosclerosis (Vascular disorders) | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 0
Flushing (Vascular disorders) | 3 | 1 | 1
Hot flush (Vascular disorders) | 0 | 2 | 0
Hypertension (Vascular disorders) | 6 | 3 | 2
Hypotension (Vascular disorders) | 3 | 1 | 1
Pallor (Vascular disorders) | 0 | 1 | 0
Thrombophlebitis (Vascular disorders) | 0 | 0 | 1
Thrombosis (Vascular disorders) | 0 | 1 | 0
Varicose vein (Vascular disorders) | 0 | 0 | 1
Enterocolitis (Gastrointestinal disorders) | 0 | 1 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Babesiosis (Infections and infestations) | 1 | 0 | 0
Oral herpes (Infections and infestations) | 2 | 0 | 0

LIMITATIONS AND CAVEATS:
Due to sponsor's business decision, the clinical trial was terminated by the sponsor.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-23): https://cdn.clinicaltrials.gov/large-docs/03/NCT02656303/Prot_SAP_000.pdf